CLINICAL TRIAL: NCT05956509
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Efficacy, and Tolerability of ABBV-950 for the Treatment of Upper Limb Spasticity in Adult Post-Stroke Patients
Brief Title: Study of Intramuscular Injections of ABBV-950 to Assess Adverse Events and Change in Disease Activity in Adult Participants With Upper Limb Spasticity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-499
Record Dates: First submitted 2023-07-14; First posted 2023-07-21 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Upper Limb Spasticity
Keywords: Spasticity; Upper Limb Spasticity; Stroke; ABBV-950; Botulinum toxin type A
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- Part 1: ABBV-950 Dose A (Experimental): Participants will receive ABBV-Dose A on Day 1.
  Interventions: Biological: ABBV-950
- Part 1: Placebo for ABBV-950 Dose A (Placebo Comparator): Participants will receive placebo for ABBV-950 on Day 1.
  Interventions: Drug: Placebo for ABBV-950
- Part 1: ABBV-950 Dose B (Experimental): Participants will receive ABBV-950 Dose B on Day 1.
  Interventions: Biological: ABBV-950
- Part 1: Placebo for ABBV-950 Dose B (Placebo Comparator): Participants will receive placebo for ABBV-950 on Day 1.
  Interventions: Drug: Placebo for ABBV-950
- Part 1: ABBV-950 Dose C (Experimental): Participants will receive ABBV-950 Dose C on Day 1.
  Interventions: Biological: ABBV-950
- Part 1: Placebo for ABBV-950 Dose C (Placebo Comparator): Participants will receive placebo for ABBV-950 on Day 1.
  Interventions: Drug: Placebo for ABBV-950
- Part 2: BOTOX Dose A (Active Comparator): Participants will receive BOTOX Dose A on Day 1.
  Interventions: Biological: BOTOX
- Part 2: ABBV-950 Dose A (Experimental): Participants will receive ABBV-950 Dose A on Day 1.
  Interventions: Biological: ABBV-950
- Part 2: ABBV-950 Dose B (Experimental): Participants will receive ABBV-950 Dose B on Day 1.
  Interventions: Biological: ABBV-950
- Part 2: ABBV-950 Dose C (Experimental): Participants will receive ABBV-950 Dose C on Day 1.
  Interventions: Biological: ABBV-950
- Part 2: Placebo for ABBV-950 (Placebo Comparator): Participants will receive placebo for ABBV-950 on Day 1.
  Interventions: Drug: Placebo for ABBV-950

INTERVENTIONS:
Biological: ABBV-950 — Intramuscular (IM) Injection
  Other Names: Botulinum toxin type A
  Arms: Part 1: ABBV-950 Dose A; Part 1: ABBV-950 Dose B; Part 1: ABBV-950 Dose C; Part 2: ABBV-950 Dose A; Part 2: ABBV-950 Dose B; Part 2: ABBV-950 Dose C
Biological: BOTOX — Intramuscular (IM) Injection
  Other Names: OnabotulinumtoxinA
  Arms: Part 2: BOTOX Dose A
Drug: Placebo for ABBV-950 — Intramuscular (IM) Injection
  Arms: Part 1: Placebo for ABBV-950 Dose A; Part 1: Placebo for ABBV-950 Dose B; Part 1: Placebo for ABBV-950 Dose C; Part 2: Placebo for ABBV-950

SUMMARY:
Spasticity is often observed as muscle tightness and stiffness in the upper and/or lower limbs. Upper limb spasticity can interfere with joint movement and its severity can range from mild to severe. Common causes of spasticity include cerebral palsy, traumatic brain injury, multiple sclerosis, spinal cord injury, and stroke. This study will assess how safe and effective ABBV-950 is in treating upper limb spasticity in adult post-stroke participants. Adverse events and change in symptoms will be assessed.

ABBV-950 in an investigational drug being developed for treating spasticity. This study is conducted in 2 parts. In Part 1, participants are assigned to receive different doses of ABBV-950 or placebo. There is 1 in 4 chance that participants will be assigned to receive placebo. In Part 2, participants will be randomly assigned to receive BOTOX, ABBV-950, or placebo. There is 1 in 5 chance for participants to receive placebo. Approximately 297 adult post-stroke participants with upper limb spasticity will be enrolled at approximately 50 sites in the United States.

In Part 1, participants will receive intramuscular (IM) injections of ABBV-950 or placebo on Day 1. In Part 2, participants will receive IM injections of BOTOX, ABBV-950, or placebo on Day 1. All participants will be followed for 24 weeks.

There may be higher treatment burden for participants in this trial compared to the standard of care. Participants will attend regular clinic visits during the study. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of upper limb spasticity due to stroke, with most recent stroke occurring at least 12 weeks prior to the Screening visit.
* Modified Ashworth Scale-Bohannon (MAS-B) score of >= 3 in the wrist flexors, and a score of >= 1+ in the finger flexors and MAS-B score of >= 2 elbow flexors at both Screening and Visit 2 (Baseline).

Exclusion Criteria:

* Additional strokes in the 12 weeks preceding the most recent stroke and in the opinion of the investigator, is not at significant risk of experiencing another stroke during the study period.
* Spasticity in the contralateral upper limb that requires treatment.
* Presence of fixed contractures in muscles of wrist, elbow, fingers.
* Botulinum toxin treatment of any serotype in the 20 weeks prior to Day for upper limb spasticity and in the 12 weeks prior to Day 1 for any indication other than upper limb spasticity.
* Previous surgical intervention, nerve block, or muscle block for the treatment of spasticity in the study limb in the last 12 months.
* Injection of corticosteroids or anesthetics in the study limb within 12 weeks.
* Casting of the upper limbs within 12 weeks.
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, and/or amyotrophic lateral sclerosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Wrist Modified Ashworth Scale-Bohannon (MAS-B) | Up to Week 6
  MAS-B measures muscle tone based on grading the resistance encountered in a specific muscle group by means of passively moving a limb through its range of motion at a study-specified velocity. Score ranges from 0 (No increase in muscle tone) through 4 (Affected part(s) rigid in flexion or extension).
Number of Participants Experiencing Adverse Events | Up to Week 24
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

SECONDARY OUTCOMES:
Change in Clinician Global Impression of Change (CGI-C) Score | Up to Week 6
  CGI-C is a 9-point rating scale used to measure the clinician's impression of overall treatment response since the first dose of study intervention. CGI-C scores range from -4 = very marked worsening to +4 = very marked improvement.
Change in Clinician Global Impression of Severity (CGI-S) Score | Up to Week 6
  CGI-S is a 5-point rating scale used to measure the clinician's or trained personnel's impression of the current severity of the participant's upper limb spasticity. Scores range from 0 = no spasticity to 4 = very severe.
Percentage of Participants Achieving Wrist MAS-B Responder Status | Up to Week 6
  MAS-B measures muscle tone based on grading the resistance encountered in a specific muscle group by means of passively moving a limb through its range of motion at a study-specified velocity. Score ranges from 0 (No increase in muscle tone) through 4 (Affected part(s) rigid in flexion or extension). Responder is defined as participant with >= 1 grade improvement from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (9):
- United States (9):
  - North County Neurology Associates /ID# 256333, Carlsbad, California
  - Rancho Los Amigos National Rehabilitation center /ID# 255335, Downey, California
  - Neuro Pain Medical Center /ID# 256036, Fresno, California
  - New England Institute for Clinical Research /ID# 255020, Stamford, Connecticut
  - MedStar National Rehabilitation Hospital /ID# 255630, Washington D.C., District of Columbia
  - JEM Research Institute /ID# 258782, Lake Worth, Florida
  - Kansas Institute of Research /ID# 254998, Overland Park, Kansas
  - University of Missouri Hospital /ID# 255310, Columbia, Missouri
  - Ut Southwestern Medical Center /Parkland Health and Hospital System /Id# 255328, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-499